CLINICAL TRIAL: NCT02296658
Title: A Phase II Trial of Intensity-Modulated Radiotherapy Combined With S-1 Based Chemotherapy in Completely Resected Gastric Cancer
Brief Title: A Phase II Study of Postoperative S-1-Based Chemoradiotherapy in Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Wang Xin, Cancer Hospital, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2013RE-088
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Stomach Neoplasms; Chemoradiotherapy, Adjuvant; Radiotherapy, Intensity-Modulated
MeSH Terms: conditions — Stomach Neoplasms | interventions — Radiotherapy, Intensity-Modulated; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- S-1 based chemoradiotherapy (Experimental): S-1,80mg/m2/d,peroral BID,in treatment days concurrently with intensity-modulated radiotherapy in a standard manner.
  Interventions: Radiation: intensity-modulated radiotherapy; Drug: S-1

INTERVENTIONS:
Radiation: intensity-modulated radiotherapy — A total irradiation dose of 45 Gy was delivered in daily 1.8-Gy fractions (5 days a week over 5 weeks) to all patients.
Drug: S-1 — S-1,80mg/m2/d,peroral BID,in treatment days concurrently with intensity-modulated radiotherapy.

SUMMARY:
The aim of this phase II trial was to evaluate the feasibility, efficacy and tolerability of intensity-modulated radiotherapy combined with S-1 based chemotherapy in patients with pathologically positive lymph node after completely resected gastric cancer. Furthermore, the investigators sought to compare the dosimetric differences between the volumetric-modulated arc therapy (VMAT), Tomotherapy and intensity-modulated radiotherapy (IMRT) techniques in treatment planning for gastric cancer as adjuvant radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven positive lymph node gastric adenocarcinoma in patients undergoing R0 resection
* Any prior chemotherapy is allowed in this protocol
* No distant metastasis in liver,lung,,bone,central nervous system(CNS),no peritoneal transplantation
* No prior abdominal or pelvic radiotherapy
* Karnofsky performance status(KPS)≥ 70, predictive life span no less than 6 months
* Patients must have normal organ and marrow function as defined below:

  * Leukocytes greater than or equal to 3,000 G/L
  * Platelets: greater than or equal to 100,000/mm3
  * Hemoglobin:greater than or equal to 10g/L
  * Total bilirubin: within normal institutional limits
  * AST/ALT: less than or equal to 1.5 times the upper limit
  * Creatinine within normal upper limits
* Informed consent

Exclusion Criteria:

* Patients with other cancer history except cervical carcinoma in situ and non-malignant melanoma skin cancer
* With any distant metastasis in liver,lung,,bone,CNS,or peritoneal transplantation
* History of allergic reactions attributed to similar chemical or biologic complex to S-1
* Uncontrolled illness including, but not limited to, active infection, symptomatic heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness
* History of myocardial infarction within the past 6 months or history of ventricular arrhythmia
* History of prior radiation to the abdomen
* Pregnant or lactating females

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 3 years
Locoregional recurrence free survival | 3 years
Overall survival | 3 years
Distant metastasis free survival | 3 years

SECONDARY OUTCOMES:
Chemoradiotherapy-induced toxicities assessed by CTCAE 4.0 | during treatment and within the first 30 days after completion of chemoradiotherapy

OTHER OUTCOMES:
Comparison of dosimetric differences between radiation techniques | 1 year
  To compare the dosimetric differences between the volumetric-modulated arc therapy (VMAT), Tomotherapy and intensity-modulated radiotherapy (IMRT) techniques in treatment planning.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, Cancer Hospital, Chinese Academy of Medical Sciences (CAMS) and Peking Union Medical College (PUMC), Beijing, China